CLINICAL TRIAL: NCT02105298
Title: Effect of Volume and Type of Fluid on Postoperative Incidence of Respiratory Complications and Outcome (CRC-Study)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, M.D., Ph.D., Massachusetts General Hospital
Other Study IDs: 2013P001704; 222302 (Other Grant/Funding Number: 222302)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Failure; Acute Respiratory Failure Requiring Reintubation; Pulmonary Edema; Pneumonia; Hypoxia; Acute Kidney Injury
Keywords: Fluids; Intraoperative; Respiratory; Outcomes; Surgery; Anesthesia
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Edema; Pneumonia; Hypoxia; Acute Kidney Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Intraoperative intravenous fluid management practice varies greatly between anesthesiologists. Postoperative fluid based weight gain is associated with major morbidity. Postoperative respiratory complications are associated with increased morbidity, mortality and hospital costs. The literature shows conflicting data regarding intraoperative fluid resuscitation volume. No large-scale studies have focused on intraoperative fluid management and postoperative respiratory dysfunction.

Hypotheses:

Primary - Liberal intraoperative fluid resuscitation is associated with an increased risk of 30 day mortality Secondary - Liberal intraoperative fluid resuscitation is associated with increased likelihood of postoperative respiratory failure, pulmonary edema, reintubation, atelectasis, acute kidney injury and peri-extubation oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 upwards
* Tracheally intubated at the beginning of the procedure and extubated at the end of the procedure

Exclusion Criteria:

* Cases where the subject had additional surgeries within the previous four weeks
* Ages under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All surgical patients aged 18 upwards receiving general anesthesia at Massachusetts General Hospital between January 2007 and November 2012
Sampling Method: Probability Sample
Enrollment: 104000 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mortality | within 30 days after surgery
  Mortality within 30 days of surgery

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 3 days after surgery
  The incidence of a diagnosis of pneumonia, respiratory failure, atelectasis or pulmonary edema within 3 days after extubation in the operating room. Cases where these diagnoses were present on the day before surgery were not counted.
Acute Kidney Injury | within 48 hours of surgery
  A Creatinine increase of >0.3mg/dl or 50% from baseline (Creatinine value closest recorded to surgery but within 30 days of surgery) to maximum value measured within 48 hours postoperatively or an ICD-9 diagnosis of AKI within 7 days of surgery but not within 30 days prior to surgery
Post-extubation oxygen desaturation | within the first 10 minutes after extubation
  One or more minutes with a blood oxygen saturation below 90% during the first ten minutes after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Eikermann, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States